CLINICAL TRIAL: NCT00343096
Title: Buccal, Intranasal or Intravenous Lorazepam for the Treatment of Acute Convulsions in Children in Blantyre, Malawi: a Randomized Trial
Brief Title: Randomized Trial Comparing 3 Routes of Delivering Lorazepam to Children.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The buccal arm of the study was 30% less effective in stopping seizures within 10 minutes compared with the IV dose. This met a stopping rule for the study
Sponsor: Kamuzu University of Health Sciences (Other)
Responsible Party: Principal Investigator, Elizabeth Molyneux, Professor of Paediatircs, Kamuzu University of Health Sciences
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: The BIVIN Trial
Record Dates: First submitted 2006-06-21; First posted 2006-06-22 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Status Epilepticus; Convulsions
Keywords: intranasal; buccal; lorazepam; paediatric; convulsions
MeSH Terms: conditions — Status Epilepticus; Seizures | interventions — Lorazepam

INTERVENTIONS:
Drug: Lorazepam — All doses 0.1mg/kg once, repeat after 10 minutes x1

SUMMARY:
This study aims to address the hypothesis that Lorazepam (an anticonvulsant) is as effective when given via the intranasal or buccal route as the intravenous route in terminating convulsions in children.

DETAILED DESCRIPTION:
Convulsions are common in children. Prompt treatment with an effective anticonvulsant reduces longterm morbidity and mortality. The use of intravenous lorazepam as first line therapy in acute childhood convulsions where venous access has been obtained is widely accepted in developed countries. However, intravenous access can be a problem out of hospital or in small children.

Benzodiazepines such as Lorazepam have long been the mainstay of first line therapy for acute convulsions but there is insufficient clinical evidence as to the optimal mode of administration when venous access has failed. Lorazepam can be given via the intranasal and buccal route offering the potential to be as effective as intravenous lorazepam whilst being easier to administer and avoiding the need for intravenous cannulation.

To date there are no large published studies that have evaluated the efficacy and safety of intranasal or buccal lorazepam compared to intravenous lorazepam in the treatment of acute convulsions. In this study we wish to address the urgent need to obtain randomized controlled data in treating acute convulsions in children using a drug and delivery system that is safe, effective and easy to use in our setting.

ELIGIBILITY:
Inclusion Criteria:

children with acute generalized seizures, continuing for a minimum of 5 minutes, who have not received any anti-convulsant therapy within 1 hour of presentation.

Exclusion Criteria:

Children who have received anticonvulsant treatment within 1 hour prior to assessment. Any child whose seizures cease following correction of hypoglycaemia. Children with a known adverse reaction to lorazepam.

Ages: 2 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2006-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Whether cessation of fit was achieved within ten minutes or not.

SECONDARY OUTCOMES:
Frequency of additional drugs required to terminate presenting seizure
Frequency of cardio-respiratory side effects
Seizure recurrence within 24 hours of terminating the presenting seizure
Time from identification of a fitting child to cessation of fit.
Outcome of patients including any neurological sequelae at hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Molyneux, Principal Investigator — College of Medicine
Locations (1):
- Queen Elizabeth Central Hospital, Paediatric Dept, Box 360, Blantyre, Malawi